CLINICAL TRIAL: NCT05028647
Title: Validazione di un Supporto Tecnologico Educativo Per Ragazzi Con Dislessia. Studio Aperto Randomizzato e Controllato
Brief Title: VAlidation of an Educational Technological Tool for Dyslexic Adolescents: an Open Controlled Study
Acronym: FORDYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Universidad de Burgos (Other); Asociatia Bucuresti Pentru Copii Dislexici (Unknown); Augumented Reality Software ARSOFT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 823
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Dyslexia
Keywords: learning disability
MeSH Terms: conditions — Dyslexia; Learning Disabilities

STUDY DESIGN:
Intervention Model Description: open randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VR treatment (Active Comparator): 5 subjects per country aged 13-16 treated with VR supported (Oculos) program, one hour a day for 5 days
  Interventions: Device: Virtual reality training
- AR treatment (Active Comparator): 5 subjects per country aged 10-13 treated with AR supported (tablet) program, one hour a day for 5 days
  Interventions: Device: Augmented reality training
- control age 13-16 (No Intervention): dyslexic subjects aged 13-16 not randomized to active treatment
- Control age 10-12 (No Intervention): dyslexic subjects aged 10-12 not randomized to active treatment

INTERVENTIONS:
Device: Virtual reality training — one hour a day for 5 days of engagement in tasks proposed by a specially crafted software through a VR device (Oculos)
  Arms: VR treatment
Device: Augmented reality training — one hour a day for 5 days of engagement in tasks proposed by a specially crafted software through a AR device (tablet)
  Arms: AR treatment

SUMMARY:
Virtual reality (VR) and augmented reality (AR) are gaining importance in the rehabilitation programs for learning disabilities. The project will test tolerability and efficacy of a VR/AR specially developed tool to improve reading abilities of adolescents with dyslexia aged 10-16

DETAILED DESCRIPTION:
Dyslexia is the most common form of learning difficulty, with a prevalence of at least 10 percent, putting more than 700 million children and adults worldwide at risk of life-long illiteracy and social exclusion (Springer-Charolles, Siegel, Jiménez & Ziegler, 2011). In the EU context 2,500,000 dyslexic school children in the EU have a specific disorder in learning to read and spell (dyslexia). Dyslexia is one of the development disorders that has been most discussed and researched, however, intervention through technology is relatively recent. The wide repertoire of manifestations and problems associated with dyslexia can be an obstacle to access to a standardized curriculum. It can also make it difficult to access the training or mobility programs provided by the European Union.

The FORDYS-VAR main objective is to provide an opportunity to improve the learning of people with dyslexia through technology, specifically Virtual Reality (VR) and Augmented Reality (AR). Introducing these technologies in the process of evaluation and intervention can become a key element to improve the effectiveness of learning and the improvement of their training experience.

Working with the AR and the VR provides people with dyslexia a safe and controlled environment, improves their motivation, contributes to generate high levels of interaction. Another advantage that we must emphasize is that you get an immediate feedback through technology, which contributes to improve visual skills and memory.

The transnationally approach of this project is needed because dyslexia occurs in all languages. Also we must consider that depending on the language, dyslexia will manifest itself in different ways. Target groups: (1) Children with dyslexia that will be the end-users of the materials developed; (2) Professionals involving in providing formal and non-formal treatment of dyslexia: Therapist, educators; (3) Families of dyslexic children.

The FORDYS-VAR project aims to be a reference in the definitive treatment of dyslexia, The creation of VR and AR materials for improvement the treatment of dyslexia in school children will be the final goal of the project. As mentioned before, "the definitive treatment" has not yet been found, but what is known is that the best treatments or the most effective include aspects such as intensive sessions, explicit instructions, individual or small group work and special attention must be paid to the phonological awareness and compensation strategies. It has also been seen that in many cases the adherence to treatments is not very high since they tend to be very repetitive and not very stimulating (children end up being bored). Currently, the applied treatments are multisensory structured language education (MSLE). They are usually multisensory, highly structured and sequential. For this reason, VR and AR fit perfectly into improving the efficacy of these treatments.

* VR and AR will be immersive and interactive. That is, not only glasses will be used to see, but also proposed tools will promote the interaction with gestural recognition so that the experience is more immersive and, therefore, more active (this will impact in the interaction with gestural recognition so that the experience is more immersive and, therefore, more active (child engagement). Furthermore, a classroom (or a more playful environment) will be simulated in which there will be different objects with which the school children can interact, for example a blackboard, and a desk with a notebook.
* For the creation of the catalog of objects to work with AR, it will be directed above all to work in the classroom and at home with the parents aimed at the building students' phonological awareness and increasing their level of vocabulary.

A participatory design (co-design) for the development of VR materials from the experiences / needs of the users will be employed in building the programs to be run on VR (Oculos) or AR (tablets) apparatus.

A social impact assessment of the activities and results implemented by the project which will take into account gender issues.

20 dyslexic boys and girls will be recruited in each country (60 total). Half of them will be in the age group of 10-12y and half 13-16y.

All recruited subjects will complete the PIRLS questionnaire at admission. 5 subjects for each age group will be randomly allocated to the intervention arm by a PC generated randomization list and will be exposed to the VR (subjects aged 13-16) or AR (subjects aged 10-12) treatment. The treatment will last one week and imply 1 hour each day of supervised use of the devices loaded with the specially developed software. At the end of the training week the participants will repeat the PIRLS questionnaire and will complete the Technology acceptance questionnaire and the Technical aspects questionnaire (both validated tools) to assess the tolerability of the treatment. The group of subjects not exposed to treatment will repeat the PIRLS questionnaire after one month.

The results of the tolerability questionnaires will be analysed to assess safety and acceptance of the tools, while the possible difference in the PIRLS score pre/post treatment will give information on efficacy.

ELIGIBILITY:
Inclusion Criteria:

* junior high school students aged 10-16y
* diagnosis of dyslexia

Exclusion Criteria:

* cognitive impairment (QI<85),
* diagnosis of conditions not compatible with the exposure to VR or AR environments:
* epilepsy,
* photosensibility,
* vestibular problems,
* perceptual problems,
* psychiatric conditions)

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
scores at the TAM (technology assessment questionnaire) | 5 days
  tolerability on the validated scale scoring 20-100 (higher score better acceptance)

SECONDARY OUTCOMES:
change in the PIRLS (Proficiency in reading skills) questionnaire scores | 5 days
  efficacy. scoring is qualitative on the various items reflecting the reading proficiency, typical scores between 300-700 (higher score better performance)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Medea, Conegliano, Treviso, Italy

IPD SHARING:
Plan to Share IPD: Undecided